CLINICAL TRIAL: NCT00547846
Title: A Phase II Clinical Study of PDC-748 in Patients With Acute Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: PH-CP013; SBIR: 2Z950430
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Acute Cough
Keywords: Cough; Antitussive; PDC-748; PhytoHealth
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PDC-748

SUMMARY:
The pharmacological effects of PDC-748 were tested in numerous in vitro and in vivo studies. The existing pharmacologic findings suggest that PDC-748 possesses certain inhibitory activity to the citric acid- and capsaicin-induced cough reflex in guinea pigs with a dose-dependent manner. Furthermore, a previous Phase I/II uncontrolled, dose-escalating study has shown PDC-748 to be well tolerated and may help to alleviate daytime cough with a dose-responding manner.Hence, PhytoHealth Corporation intends to carry out a Phase II investigation to confirm the preliminary findings using placebo in the comparator group, and to further investigate PDC-748 with a dose escalating manner to establish the dose-response range for its antitussive effect, and if possible, to determine the maximal tolerable dose of PDC-748.

This is a randomized, double-blind, placebo-controlled, dose escalating study to evaluate the safety and efficacy of the escalating dose levels of PDC-748 in patients with acute cough.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute cough ;
* Men or women aged ≥ 20 years old;
* Patients with Cough Symptom Score(daytime) between 2 and 4, inclusively;
* Patients are willing and able to comply with the study procedures and sign the informed consent.

Exclusion Criteria:

* Patients with chronic cough ;
* Patients with chronic airway disease;
* Patients with respiratory tract malignancy;
* Patients with clinically suspected low respiratory tract infection;
* Patients with abnormal liver or kidney functions
* Patients taking antitussives, sleeping pills, sedative medications, or herbal products;
* Pregnant or breastfeeding patients; female patients of child bearing potential who do not agree to practice effective birth control;
* Patient's symptom of acute cough may be due to heart failure or may be induced by other medications such as ACE inhibitor medications, as determined by the investigator;
* Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with the assessments of safety or efficacy during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, or hematological disease as determined by the clinical judgment of the investigator;
* Use of any investigational drug or participation of any clinical trial within 28 days prior to this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Huang Tsai, M.D., Principal Investigator — Chang Gung Memorial Hospital; Ying Huang Tsai, PI, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang-Gung Memorial Hospital,Taiwan, Taipei City/ Taoyuan County, Taiwan,ROC, Taiwan